CLINICAL TRIAL: NCT04651140
Title: Research on the Effect and Mechanism of Aerobic Exercise on Parkinson's
Brief Title: Research on the Effect and Mechanism of Aerobic Exercise on PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zhang Ying, Professor, The First Hospital of Jilin University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zhang Ying
Record Dates: First submitted 2020-11-08; First posted 2020-12-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-11

CONDITIONS: Parkinson's Disease; Physical Exercise
Keywords: Parkinson's Disease; Physical exercise; Mechanism
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tremor group (Active Comparator): Participants in the tremor group have tremor as the main clinical manifestation
  Interventions: Behavioral: aerobic exercise
- Stiff group (Active Comparator): Participants in the tremor group have stiff as the main clinical manifestation
  Interventions: Behavioral: aerobic exercise

INTERVENTIONS:
Behavioral: aerobic exercise — Participants ride an Acon-8650 model exercise bicycle 3 times a week for 1 hour each time for four consecutive weeks

SUMMARY:
This trial is expected to recruit patients with primary Parkinson's disease and give them four consecutive weeks of aerobic exercise to observe its effect on Parkinson's disease and explore its mechanism

DETAILED DESCRIPTION:
This trial is expected to recruit patients with primary Parkinson's disease who are distributed into tremor group and stiff group and give them the same kind of four consecutive weeks of aerobic exercise to observe its effect on Parkinson's disease and explore its mechanism

ELIGIBILITY:
Inclusion Criteria:

* Participants were diagnosed primary PD according to the 2015 MDS diagnostic criteria
* Participants are between 55 and 65 years old

Exclusion Criteria:

* Severe heart
* liver dysfunction
* kidney dysfunction
* severe cognitive dysfunction
* severe anxiety and depression
* history of mental illness
* history of cerebral infarction or ischemic attack in the past three months
* acute myocardial infarction or acute coronary in the past three months
* Parkinson's Pulse syndrome
* medication history (drugs that improve blood circulation in the brain and increase the excitability of the nervous system)

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-United Parkinson's Disease Rating Scale (MDS-UPDRS) | changes of MDS-UPDRS score from baseline at four weeks
  to assess the motor and nonmotor function of PD,0-200 scores,the higher scores mean lower function
Montreal Cognitive Assessing(MoCA) score | changes of MoCA score from baseline at four weeks
  to assess the cognitive function of PD,0-30 scores,the higher scores mean better function
The Epworth Sleeping Scale(ESS) | changes of ESS score from baseline at four weeks
  to assess the degree of drowsiness, 0-24 scores, the higher scores mean severe drowsiness
Non-Motor Symptom Scale (NMSS) | changes of NMSS score from baseline at four weeks
  to assess the non-motor of PD , 0-120 scores, the higher scores mean severe non-motor damage

SECONDARY OUTCOMES:
cerebral blood variation by Head MRI | changes of the cerebral blood from baseline at four weeks
  to assess the cerebral blood variation by head MRI
cerebral blood flow velocity | changes of the cerebral blood flow velocity from baseline at four weeks
  cerebral blood flow velocity is recorded using transcranial Doppler and a servo-controlled plethysmograph respectively.
the level of arterial blood pressure | changes of the arterial blood pressure from baseline at four weeks
  arterial blood pressure is recorded using transcranial Doppler and a servo-controlled plethysmograph respectively. Both systolic and diastolic pressures will be assessed during the study period.
the concentration of microRNA in peripheral blood by gene chip | changes of microRNA from baseline at four weeks
  to test the the concentration of microRNA in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhang, Doctor, Study Director — The First Hospital of Jilin University
Locations (1):
- FirstJilinU, Changchun, China

IPD SHARING:
Plan to Share IPD: No